CLINICAL TRIAL: NCT01180166
Title: Phase II Study of Nimotuzumab and Concurrent Radiotherapy and Capecitabine for Inoperable Locally Advanced or Recurrent Gastric Cancer
Brief Title: Combination of Nimotuzumab,Capecitabine and Radiotherapy for Inoperable or Recurrent Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., vice chair of radiation department, Chinese Academy of Medical Sciences, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-010
Record Dates: First submitted 2010-08-03; First posted 2010-08-12 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Gastric Cancer; Concurrent Chemoradiotherapy
Keywords: Gastric cancer; concurrent chemoradiotherapy; target therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nimotuzumab (Experimental): Combination of nimotuzumab and capecitabine concurrent chemoradiotherapy is received by patients.
  Interventions: Drug: nimotuzumab

INTERVENTIONS:
Drug: nimotuzumab — 200 milligram (mg) of nimotuzumab per week during radiation period
  Other Names: Nimotuzumab injection, Tai Xin-sheng

SUMMARY:
The prognosis of patients with inoperable locally advanced or residual/relapsed gastric cancer is rather poor. Concurrent capecitabine chemoradiotherapy is safe and recommended. Nimotuzumab, an anti-EGFR (epidermal growth factor receptor) monoclonal antibody, has shown its antitumor safety and efficiency in many phase I/II studies. Efficiency of combination of these treatment need to be further analyzed.

DETAILED DESCRIPTION:
There is no standard treatment for patients with inoperable locally advanced or residual/relapsed gastric cancer. For the former ones, 5-fluorouracil(5-FU) based concurrent chemoradiotherapy is a recommended treatment regimen. Concurrent capecitabine chemoradiotherapy showed similar results. So far, more and more studies have shown that drugs targeting at EGFRs play an important role in antitumor treatment. Nimotuzumab, an anti-EGFR monoclonal antibody, has shown its safety and efficiency in many phase I/II studies. Because of poor survival of patients with inoperable locally advanced or residual/relapsed gastric cancer, the efficiency of nimotuzumab plus concurrent capecitabine chemoradiotherapy need to be further analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, male or female
* Gastric cancer with measurable lesions, and the diameter is at least 1 cm
* Karnofsky score: at least 70
* Estimated survival: at least 6 months
* No prior target therapy or radiotherapy
* No severe hypertension, cardiac disease, or diabetes mellitus
* Normal blood routine and chemical tests
* Signed consent

Exclusion Criteria:

* Other malignancies simultaneously except in situ cervix or non-melanoma skin cancer
* Extensive distant metastases
* Pregnancy or in lactation
* Allergic to 5-Fluorouracil

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 1 year progression-free survival
  progression-free survival: the time between tumor regression to progression

SECONDARY OUTCOMES:
overall responses | 1 month after treatment
  the overall responses: complete response (CR)+ partial response(PR)+ stable disease (SD) rates based on World Health Organization(WHO) evaluation system
overall survival time | 1 month after treatment
  median overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: jing jin, M.D., Principal Investigator — Chinese Acedemy of Medical Sciences
Locations (1):
- Radiotherapy Department of Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China